CLINICAL TRIAL: NCT06109168
Title: Correlation of SpO2/FIO2 Ration With PaO2/FIO2 Ratio in Acute Respiratory Distress Syndrome (ARDS) Patients in the ICU of H. Adam Malik Hospital
Brief Title: Correlation of SpO2/FIO2 Ratio With PaO2/FIO2 Ratio in ARDS Patients in the ICU of H. Adam Malik Hospital
Acronym: MNO
Status: Completed | Type: Observational
Sponsor: RS H Adam Malik (Other)
Responsible Party: Principal Investigator, Agus pramono, Resident of Department of Anesthesiology and Emergency Medicine of Medical Faculty USU, RS H Adam Malik
Other Study IDs: 536/KEPK/USU/2023
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Ards
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood Gas Analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study to apprehend the relation of SpO2/FiO2 to PaO2/FiO2 in ARDS patients.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is a life-threatening condition that requires immediate treatment. The measurement of the PaO2/FiO2 (P/F) ratio is the main choice for assessing the severity of ARDS with an invasive method that requires arterial blood gas (ABG) analysis. This study was conducted to determine the relationship between the SpO2/FiO2 ratio and the PaO2/FiO2 ratio in ARDS patients at HAM General Hospital. This observational study used a cross-sectional research method with the total sample of 29 intubated ICU patients diagnosed with ARDS. Patients with congestive heart failure, anemia, and systolic blood pressure <90 mmHg were excluded from the study. The results of this study showed a positive correlation between the PaO2/FiO2 and SpO2/FiO2 ratios with a correlation coefficient of 0.955 and a p-value of 0.001. There was a relationship between the S/F ratio and the P/F ratio in assessing the severity of ARDS with a p-value of <0.05. This study shows that the SpO2/FiO2 (S/F) ratio has a good correlation with the PaO2/FiO2 (P/F) ratio in patients with ARDS, so it can be used as a predictor of ARDS and can be beneficial in clinical practice. It should be noted that the SpO2/FiO2 ratio has several factors that can affect its accuracy, so careful assessment is needed.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patient
* intubarted patient

Exclusion Criteria:

* Cardiac congenital disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intubated patients in ICU
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation of SpO2/FIO2 Ratio with PaO2/FIO2 Ratio in Acute Respiratory Distress Syndrome (ARDS) Patiens in the ICU of H. Adam Malik Hospital | June - August 2023
  ICU patients

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP H. ADam Malik, Medan, North Sumatra, Indonesia